CLINICAL TRIAL: NCT00330577
Title: 24-Hour Intraocular Pressure (IOP) And Blood Pressure Control In Glaucoma And Ocular Hypertension Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A594
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost; Lubricant Eye Drops

INTERVENTIONS:
Drug: timolol maleate 0.5%
Drug: latanoprost/timolol fixed combination
Drug: placebo (artificial tears)

SUMMARY:
The purpose of this study is to compare the short-term mean 24-hour intraocular pressure control, 24-hour blood pressure effect and safety of Latanoprost/Timolol fixed combination given once in the evening with placebo once in the morning versus timolol maleate 0.5% given twice daily in patients with ocular hypertension and primary open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* POAG
* OHT

Exclusion Criteria:

* Advanced glaucoma
* Arterial Hypertension

Ages: 29 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AGP Konstas, MD, PhD, Principal Investigator — Glaucoma Unit, A University Dept of Ophthalmology, AHEPA Hospital
Locations (1):
- Glaucoma Unit, A University Dept of Ophthalmology, AHEPA Hospital, Thessaloniki, Greece